CLINICAL TRIAL: NCT00281905
Title: Management of Children Aged Less Than 3 Years With Brain Tumors
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Children With Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454575; CCLG-CNS-9204; EU-20574; CCLG-CNS-1992-04
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-06

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma
Keywords: untreated childhood brain stem glioma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; untreated childhood cerebellar astrocytoma; childhood choroid plexus tumor; childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma; untreated childhood medulloblastoma; childhood oligodendroglioma; untreated childhood supratentorial primitive neuroectodermal tumor; disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Astrocytoma; Choroid Plexus Neoplasms; Oligodendroglioma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Methotrexate; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: methotrexate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after chemotherapy may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with or without radiation therapy works in treating children with brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in children under 36 months of age with primary brain or brain stem tumors treated with vincristine, methotrexate, carboplatin, cyclophosphamide, and cisplatin with or without radiotherapy.
* Determine the event-free survival and overall survival in children treated with this regimen.
* Determine the pattern of local recurrence or occurrence of CNS metastases in children treated with this regimen.
* Determine the quality of life in children treated with this regimen.
* Determine the tolerability and long-term toxicity of this regimen in these children.
* Determine the proportion of children who require radiotherapy after treatment with this regimen.
* Determine the prognosis of children who receive both chemotherapy and radiotherapy.
* Determine the nature and behavior of brain tumors in very young children.

OUTLINE: This is a multicenter study.

* Chemotherapy: Patients receive vincristine IV on days 0, 14, and 28; carboplatin IV over 4 hours on day 0; methotrexate IV continuously over 24 hours on day 14; cyclophosphamide IV over 4 hours on day 28; and cisplatin IV continuously over 48 hours on days 42 and 43. Courses repeat every 56 days (8 weeks) for up to 12 months. Patients who achieve a complete response proceed to observation, as do those achieving a partial response with no tumor present on biopsy. Patients with biopsy proven residual tumors after 12 months of chemotherapy or recurrent tumors that don't have the potential to spread through the cerebrospinal fluid (CSF) proceed to local radiotherapy. Patients with unresponsive disease or progressive disease that has the potential to spread through the CSF proceed to craniospinal radiotherapy.
* Local radiotherapy: Patients undergo local radiotherapy 5 days a week for 5-5½ weeks.
* Craniospinal radiotherapy: Patients undergo craniospinal radiotherapy 5 days a week for 4 weeks.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed periodically for at least 2 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Brain stem tumor (histological confirmation not required)
  * Histologically confirmed primary intracranial brain tumor of 1 of the following histologies:

    * Anaplastic (malignant) astrocytoma
    * Glioblastoma
    * Anaplastic (malignant) oligodendroglioma
    * Ependymoma
    * Anaplastic (malignant) ependymoma
    * Anaplastic (malignant) oligoastrocytoma
    * Choroid plexus carcinoma
    * Astroblastoma
    * Polar spongioblastoma
    * Gliomatosis cerebri
    * Anaplastic (malignant) ganglioglioma
    * Pineoblastoma
    * Mixed pineocytoma or pineoblastoma
    * Medulloepithelioma
    * Neuroblastoma
    * Ependymoblastoma
    * Primitive neuroectodermal tumors (PNETs), including medulloblastoma or cerebral or spinal PNETs
* Has undergone surgery or biopsy of the tumor within the past 2-4 weeks

PATIENT CHARACTERISTICS:

* No concurrent unrelated disease, including hematological or renal disease, that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* Prior steroids allowed
* No concurrent steroids as anti-emetics

  * Concurrent steroids allowed for control of tumor-related symptoms

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 1992-06

PRIMARY OUTCOMES:
Response rate
Event-free survival
Local recurrence or occurrence of CNS metastases
Quality of survival
Tolerance
Long-term toxicity
Proportion of patients requiring radiotherapy
Prognosis of children who receive both chemotherapy and radiotherapy
Nature and behavior of brain tumors

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grundy, MD, PhD, Study Chair — Queen's Medical Center
Locations (21):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales